CLINICAL TRIAL: NCT03025633
Title: Explaining the Invisible - A Study to Evaluate the Effectiveness of Delivering Radiotherapy Treatment Information in a Visual Manner Using the PEARL System
Brief Title: Explaining the Invisible Using the PEARL System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HullEastYorkshireNHS
Record Dates: First submitted 2016-12-20; First posted 2017-01-19 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: PEARL
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - PEARL (Other): Group A will receive a combination of verbal and visual pre-treatment information via the use of PEARL.
  Interventions: Other: PEARL
- Group B - NON PEARL (No Intervention): Group B will receive verbal only pre-treatment information.

INTERVENTIONS:
Other: PEARL — PEARL, is a commercially available PC-based tool that provides a realistic and functional 3D model of a linac and, having uploaded example treatments it can demonstrate the treatment procedure and also relevant anatomical information.
  Arms: Group A - PEARL

SUMMARY:
Radiotherapy uses high doses of x-rays directed at tumours to kill them, an unfortunate side effect is healthy surrounding tissue will receive some of the x-ray dose and is damaged. Approximately 22% of radiotherapy patients receive treatment to cure prostate cancer. The technique used requires patients to maintain full bladder and empty bowel because they are next to the prostate, the aim of radiotherapy planning is to minimise the radiation dose received to healthy organs and tissues as this will reduce side effects. PEARL is commercial interactive PC software that shows realistic and functional 3D models of Linac's (machines that deliver radiotherapy treatment). Using PEARL it's possible to display realistic patient treatments including how an individual would be laid on a treatment couch and how the machine will move and sound during treatment. Additionally PEARL provides the opportunity to look inside the body to view internal anatomy and show where the radiotherapy treatment is directed.

Information prior to treatment in radiotherapy is normally given verbally one to one. The investigators believe this information can be more easily understood if PEARL is used in conjunction with this verbal exchange. PEARL gives visual and audio representation of the treatment experience, and demonstrates the reasons behind required preparations.

Research aim is to demonstrate patients who receive information using PEARL have greater understanding, reduced anxiety and reduced radiation dose. This will be tested using two groups of patients receiving radiotherapy to the prostate. Group A - Verbal information, Group B - Verbal information and PEARL demonstration. Data collection is via patient questionnaires and review of Cone Beam Computer Tomography (CBCT) images that are taken prior to each radiotherapy treatment as standard practice. CBCT's are used to locate the treatment area and assess bladder and bowel status and ensure all of these are suitable to deliver treatment accurately.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer of the prostate of the following staging: T1-3b, N0-1, M0.
* Clinical intention to treat using external radiotherapy based on three local departmental protocols: TP-CP-97, TP-CP-98 and TP-CP-99. These protocols dictate that the patients receive VMAT planned treatment, require a full bladder and empty rectum and require daily localisation using kV cone beam CT (CBCT).
* Patients consented to the study.

Exclusion Criteria:

* Patients who do not fulfil the inclusion criteria.
* Patients diagnosed with depression.
* Blind patients or patients with severe visual impairment.
* Patients with reduced understanding due to mental impairment.
* Patients not willing to consent to the study.
* Prisoners and young offenders.
* Patients who are unable to understand verbal explanations given in English.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Clinically significant reduction in the number of CBCT rescans due to protocol non-compliance (resulting from both rectum and bladder non-conformances). | 7 Months

SECONDARY OUTCOMES:
Statistically significant difference in bladder volume compliance between the two groups. | 7 Months
A statistically significant reduction in treatment-related anxiety in patients, to be assessed using pre-treatment questionnaires. | 7 Months
Increased understanding of patients, as perceived by them, regarding the radiotherapy treatment procedure in terms of accurate positioning and need for preparation (rectum/bladder management). | 7 Months

CONTACTS AND LOCATIONS:
Overall Officials: Victoria A Sykes, BSc (Hons), Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull and East Yorkshire Hospitals NHS Trust, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No